CLINICAL TRIAL: NCT00792155
Title: Autosomal Dominant Polycystic Kidney Disease Data Repository
Brief Title: Polycystic Kidney Disease Data Repository
Status: Recruiting | Type: Observational
Sponsor: The Rogosin Institute (Other)
Collaborators: Weill Medical College of Cornell University (Other); New York Presbyterian Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 0304006105
Record Dates: First submitted 2008-11-14; First posted 2008-11-17 (Estimated); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Polycystic Kidney Disease
Keywords: PKD
MeSH Terms: conditions — Polycystic Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Autosomal dominant polycystic kidney disease (PKD) is the most common inherited kidney disease, affecting more than 400,000 people in the U.S. and 5 million people worldwide. PKD is the 4th most common cause of kidney failure requiring dialysis and/or transplantation. Over half of all PKD patients develop kidney failure by age 60 years, although age of onset of kidney disease varies widely, even among members of the same family.

Despite the fact this is a relatively common problem, relatively few patients have been studied for a sufficient period of time to fully understand how patients are affected over the course of their lifetime. The reason for creating this repository is to collect information about PKD so that the investigators may fully understand its complications, including high blood pressure, heart attack, and stroke. This information may also aid in the development of improved treatment strategies.

DETAILED DESCRIPTION:
Visit #1:

* An initial detailed history, physical examination, and laboratory evaluation
* An extensive family history of PKD will be obtained from the patient.

Follow-up Study Visits:

- Patients will return to the outpatient facility for detailed follow-up examinations every other year after Visit 1.

ELIGIBILITY:
Inclusion Criteria:

* Any person, age 18 or older, with previously diagnosed ADPKD is eligible to participate.

Exclusion Criteria:

* Inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients enrolled in this study will have the diagnosis of autosomal dominant kidney disease. The diagnostic criteria for at-risk individuals (i.e., with a first degree family member with ADPKD) includes the presence of at least two(unilateral or bilateral) renal cysts, and two cysts in each kidney are considered sufficient for diagnosis in aged 15 to 29 years and in 30 to 59 years, respectively. In families of unknown genotype, the presence of three or more (unilateral or bilateral) renal cysts is sufficient for establishing the diagnosis in individuals aged 15 to 39 years, two or more cysts in each kidney is sufficient for individuals aged 40-59 years and four or more cysts in each kidney is required in individuals ≥60 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2002-11; Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Polycystic kidney disdease data repository | 30 years
  Polycystic kidney disease data repository

CONTACTS AND LOCATIONS:
Overall Officials: Jon Blumenfeld, MD, Principal Investigator — The Rogosin Institute
Locations (1):
- The Rogosin Institute, New York, New York, United States

REFERENCES:
- [Derived] Goel A, Shih G, Riyahi S, Jeph S, Dev H, Hu R, Romano D, Teichman K, Blumenfeld JD, Barash I, Chicos I, Rennert H, Prince MR. Deployed Deep Learning Kidney Segmentation for Polycystic Kidney Disease MRI. Radiol Artif Intell. 2022 Feb 16;4(2):e210205. doi: 10.1148/ryai.210205. eCollection 2022 Mar. PMID 35391774
- [Derived] Zhang Z, Bai H, Blumenfeld J, Ramnauth AB, Barash I, Prince M, Tan AY, Michaeel A, Liu G, Chicos I, Rennert L, Giannakopoulos S, Larbi K, Hughes S, Salvatore SP, Robinson BD, Kapur S, Rennert H. Detection of PKD1 and PKD2 Somatic Variants in Autosomal Dominant Polycystic Kidney Cyst Epithelial Cells by Whole-Genome Sequencing. J Am Soc Nephrol. 2021 Dec 1;32(12):3114-3129. doi: 10.1681/ASN.2021050690. Epub 2021 Dec 1. PMID 34716216